CLINICAL TRIAL: NCT04938089
Title: Effect of Periodontal Maintenance Therapy on Tooth Loss in Regular and Irregular Compliant Smokers and Non-Smokers: A Cohort Retrospective Analysis With a Follow-up Up to 40 Years
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Saint-Joseph University (Other)
Responsible Party: Principal Investigator, Roudy Khayat, Principal Investigator, Saint-Joseph University
Other Study IDs: USJ-2021-35
Record Dates: First submitted 2021-06-16; First posted 2021-06-24 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Periodontal Diseases; Tooth Loss; Compliance; Smoking
Keywords: Compliance; Maintenance; Non-Smokers; Smokers; Tobacco; Tooth Loss
MeSH Terms: conditions — Periodontal Diseases; Tooth Loss; Patient Compliance; Smoking | interventions — Maintenance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- ICS: Irregular compliant smoker
  Interventions: Other: Maintenance
- RCS: Regular compliant smoker
  Interventions: Other: Maintenance
- ICN: Irregular compliant non-smoker
  Interventions: Other: Maintenance
- RCN: Regular compliant non-smoker
  Interventions: Other: Maintenance

INTERVENTIONS:
Other: Maintenance — Regular compliant individual is defined in the study as a subject attending 100% of his/her recall visits with a maximum interval of 6 months. Irregular compliant individual is defined as a subject who missed at least one of the recall visits but continued to appear on an irregular basis with a maximum interval of 18 months, non-smoker individual is defined as a subject who never smoked, and lastly, smoker individual is defined as a subject who is smoking > 9 cigarettes per day.

SUMMARY:
Periodontal diseases are infections cause by dental plaque (Socransky, 1970). Risk factors are present which modify the course of disease progression. One of these risk factors is tobacco smoking, which was first evaluated by Pindborg in 1947 and later by Grossi et al. in 1995. They found that tobacco smoking was strongly associated with attachment loss, bone loss, and lastly, tooth loss. Tooth loss in one of the most visible results of periodontal disease, which negatively affects physiological and psychological patient's life. The effects of cigarette smoking on periodontal status are independent of the plaque index and oral hygiene of the patient, due to the direct influence of tobacco on periodontal tissues.

Several studies have demonstrated the effectiveness of periodontal therapy in reducing the rate of tooth loss as well as the importance of patient compliance with periodontal maintenance therapy and adequate oral hygiene practice in achieving this reduction. Compliance is the main problem faced in periodontal maintenance therapy. Low rates of compliance and patient adherence to a maintenance program was reported in the literature. Periodontal maintenance therapy can be considered a critical factor for success in controlling periodontitis and in the long-term maintenance of teeth. In addition, neglecting a regular periodontal maintenance therapy program has been associated with increased risk of reinfection and progression of periodontitis, as well as increased tooth loss. The establishment of a criteria for time interval between different supportive periodontal maintenance visits, is still controversial.

Smokers are associated with low level of compliance to prevent being constantly reminded of quitting smoking as well as the health complications associated with the habit. There is a void in the literature addressing the direct influence of compliance and adherence in periodontal maintenance therapy and its contribution to arrest periodontitis progression, minimizing tooth loss, specifically in tobacco smoking patients, whether they are regular or irregular compliant with a long term follow-up up to 40 years. On the other hand, there is moderate scientific evidence that the independent effect of smoking is associated with the occurrence of tooth loss in individuals undergoing periodontal maintenance therapy. Lastly, only very few studies reported the specific outcome of periodontal maintenance therapy on tooth loss in regular and irregular compliant smokers compared to regular and irregular compliant non-smokers.

The focused question in this study is "Does periodontal maintenance therapy affect annual tooth loss rates differently in regular and irregular compliant smokers and non-smokers?".

DETAILED DESCRIPTION:
Moderate scientific evidence that the independent effect of smoking is associated with the occurrence of tooth loss in individuals undergoing periodontal maintenance therapy. Only very few studies specifically reported the outcome of tooth loss and periodontal maintenance program in regular and irregular compliant smokers compared to regular and irregular compliant non-smokers.

The researcher will analyze the data provided by a specialized dental clinic in the field of periodontology and will divide the subjects into four groups: Group ICS (irregular compliant smoker), Group RCS (regular compliant smoker), Group ICN (irregular compliant non-smoker), and lastly, Group RCN (regular compliant non-smoker). The subjects present in the data will be randomly selected and divided into the appropriate groups with the aid of a permutation table. The researcher will not call the patient and perform a clinical examination but rather analyze the data retrospectively. Statistical data will be compared according to annual tooth loss rates and OR of tooth loss will be calculated for each group. After statistical analysis, the researcher will formulate proper concluding remarks regarding the importance of periodontal maintenance therapy on tooth loss rates in regular and irregular compliant smokers and non-smokers.

Primary objective:

Determine whether periodontal maintenance therapy decreases tooth loss in regular and irregular compliant smokers compared to regular and irregular compliant non-smokers after 40 years of follow-up.

Secondary objective:

Shed light on the importance of periodontal maintenance therapy, in its ability to reduce tooth loss, in smokers and non-smokers after 40 years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Smoker patients (> 9 cigarettes per day).
* At least 10 years of continued periodontal maintenance therapy.
* Diagnosis of generalized chronic periodontitis or gingivitis.
* Patient had undergone active periodontal therapy comprised of non-surgical and/or surgical therapy.

Exclusion Criteria:

* Patients with bisphosphonate therapy.
* Patients with chemo or radiotherapy.
* Patients with hormonal therapy.
* Patients with a history of refractory periodontitis or repeated abscess formation.
* Patients with debilitating diseases that could impair the immune system (HIV/AIDS, cancer, or autoimmune diseases).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The location and recruitment of patients was conducted from a specialized private dental clinic in periodontology.
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Tooth Loss | Up to 40 years
  Determine whether periodontal maintenance therapy affects tooth loss rates in regular and irregular compliant smokers compared to regular and irregular compliant non-smokers after 40 years of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Nadim Mokbel, Pr, Study Director — Saint-Joseph University; Roudy Khayat, Dr, Principal Investigator — Saint-Joseph University
Locations (1):
- Saint-Joseph University of Beirut, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided